CLINICAL TRIAL: NCT02498964
Title: Use of High Fidelity Simulation in Cardiac-specific Anesthesia Scenarios for Resident Education and Assessment
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: Buck-IRB 2015B0264
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Resident Education and Assessment of Difficult and High Acuity Scenarios That Focus on Cardiac Anesthesia
Keywords: cardiac anesthesia simulation,NASA task load index
MeSH Terms: interventions — Educational Status; Health Services Needs and Demand

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Teaching,education,feedback and practice sessions to help improve as needed — Group discussion,individual attention and teaching as needed,more teaching using different modalities like powerpoint and hands on experience

SUMMARY:
High fidelity simulations provide a unique opportunity for teaching and evaluation of knowledge, clinical reasoning, decision making and teamwork. We have developed a series of novel cardiac based simulations that review difficult learning objectives of cardiac anesthesiology rotation. We hypothesized that residents who have completed a rotation in cardiac anesthesiology will perceive these simulations to be both mentally challenging and a useful tool in preparing them for their subsequent clinical experience and for their anesthesiology board. For the first time, we have used the NASA Task Load Index Scale in evaluating Neuro Cognitive Workload during Cardiac Anesthesia Based simulation scenarios .Residents who have completed the cardiac rotation at least once would be assigned the task in small groups either a group of 2 or group of 3.The module consists of 3 different scenarios. The scenarios include, weaning the patient off of cardio pulmonary bypass, management of severe protamine drug reaction and acute hypotension from malfunction of the coronary graft in a simulated operating room in real time.

1. Setting up a Simulation Lab,almost similar to real cardiac operating rooms would have cardio-pulmonary bypass machine,transesophageal echocardiography images upon request,all emergency medications with various infusions pumps,defibrillator,real time monitors include EKG,SpO2,invasive arterial line,CVP,PAP,ETCO2,operating room surgical equipment,anesthesia machine with ventilator.
2. Tasks Assigned to the residents
3. Feed-back and Teaching Session
4. At the end of each session residents are encouraged to reflect upon how they performed and learning gaps that they perceived and areas that they felt needed to improve upon.
5. Feedback session would be followed by interactive teaching to reinforce the knowledge.
6. Evaluation of Hypothesis using NASA TLX Scale. Immediately following the Simulation based training, residents would be given the paper based NASA TLX scale to assess the neurocognitive workload

DETAILED DESCRIPTION:
The Ohio State University CSEAC Scenarios Content expert: Sujatha Bhandary MD The Ohio State University CSEAC 1st Scenario Development Form Scenario Name: Weaning from Cardiopulmonary Bypass Content expert: Sujatha Bhandary MD Date of Development: 8/29/14 Targeted Audience: CA-2, CA-3 anesthesia residents Simulation Platform: HPS

Synopsis of Scenario:

The purpose of this scenario is for the participant to take a thoughtful, systematic approach to weaning a patient off of cardiopulmonary bypass (CPB). Separation from cardiopulmonary bypass is a task which requires attention to multiple organ systems, communication with other members of the patient care team (i.e. surgeon, perfusionist), and a firm grasp of cardiopulmonary physiology. A small randomized controlled study of residents has previously demonstrated that simulation-based training in weaning from CPB has translated to improved clinical performance in the OR. While this task can at first be overwhelming for the trainee, high fidelity simulation provides an opportunity to practice this complex task in a safe environment.

The scenario will begin with the patient under general anesthesia and on cardiopulmonary bypass. The surgeon will have just completed an uncomplicated triple vessel CABG on a 57 year old male with 45 minutes of bypass time. When the participant takes over the case the patient will have a junctional bradycardia (rate 40) with a MAP of 50 mmHg, a temperature of 35 degrees celcius, and a SpO2 of 100%. The surgeon will announce that he is planning to remove the aortic cross clamp at which time the resident should call for their attending. The participant will be informed that their attending will not arrive and they will need to complete the task on their own. After removal of the cross clamp the patient will go into ventricular fibrillation. The participant will be responsible for recognizing the arrhythmia and treating the condition with lidocaine and defibrillation. After defibrillation the patient will go back into a junctional bradycardia which the participant will need to treat by pacing. At this point the participant will also need to begin ventilating the patient and treating underlying hyperkalemia (which will become evident upon obtaining an ABG). Failure to treat the hyperkalemia will result in refractory ventricular fibrillation. An echocardiogram (if requested) will reveal a normal appearing heart with good contractility. After pacing the patient, ventilating, and treating the underlying metabolic disturbances the patient can be successfully weaned off of CPB with a low dose epinephrine drip. At this point the scenario will end.

Learning Objectives:

1. Describe the conditions necessary before attempting to wean the patient from CPB
2. Demonstrate the steps involved in weaning the patient from CPB.
3. Communicate effectively with other members of the patient care team (i.e. perfusionist and surgeon) during weaning from CPB.
4. Recognize and treat arrhythmias and metabolic disturbances prior to weaning from CPB.

   Scenario Intro (read to learner) Your patient is a 57 year old male who is undergoing a triple vessel CABG (LIMA to LAD, saphenous to RCA, and saphenous to OM). In addition to CAD the patient has a history of type 2 DM and HLD. The surgeon has just completed the last graft with a total bypass time of 45 minutes. The procedure has been uncomplicated to this point. The patient has an arterial line, a 16 g IV, and an introducer with a PAC. The patient is on no infusions and is receiving isoflurance via the bypass machine. The patient is currently paralyzed. There is a transesophageal echocardiogram available upon request. The surgeon has placed epicardial pacing wires. Your task will be to wean the patient off of CPB.

   Facilitator briefing/ Curricular information:

   Prior to receiving hand-off and beginning the scenario the participant will be handed a sheet with the patient's pre-op history and physical already completed. All labs and imaging will be provided. The resident will have the opportunity to ask additional questions to the departing provider. The confederates in the room will include the cardiac surgeon and a perfusionist. Echocardiography will be available upon request as will arterial blood gases. The following infusions will already be in-line but not yet started: epinephrine, nitroprusside, and insulin. Other cardiac drugs (lidocaine, amiodarone, nitroglycerine, norepinephrine, vasopressin) will be drawn up and available. Epicardial wires coming from the surgical field. These can be connected to a pacing box which will provided upon request.

   Educational Learning Model

   Prerequisites: Completion of cardiac anesthesiology rotation Didactics Needs: Powerpoint presentation, debriefing room Learning Method: Experiential Debriefing Method: Guided reflection with peer feedback. Didactic content. Preparation Supporting Files

   • Patient preoperative report

   • PowerPoint presentation Roles
   * Cardiac Surgeon
   * Perfusionist Setting
   * OR
   * Patient intubated, sedated, paralyzed, on CPB

   Monitors Available to Participant • Code Cart with pacing/defibrillation pads • EKG monitoring

   • Five-lead electrocardiogram

   • Pulse-oximetry

   • Temperature probe
   * Capnography
   * Arterial catheter
   * Central venous catheter
   * Pulmonary artery catheter
   * Transesophageal Echocardiogram

   Other Equipment Required

   • Anesthesia machine that has passed the check out

   • Airway equipment on the cart including Macintosh 3 and Miller 2 blades, endotracheal tube sizes 6 and 7 with stylet and empty 10 mL syringe

   • Two prepared 1000 mL intravenous fluid bags on blood infusion lines

   • Pharmacologic agents available upon request: propofol, etomidate, ketamine, succinylcholine, vecuronium, midazolam, fentanyl, atropine, ephedrine, phenylephrine, epinephrine (in syringe and prepared in 100 mL saline bag), norepinephrine (in syringe and prepared in 100 mL saline bag), vasopressin, neostigmine, glycopyrrolate, metoprolol, esmolol,

   • Epinephrine, Nitroprusside, and Insulin drips connected to a manifold and in line with the patient's CVC

   • Yankauer suction

   • Record keeping material (computer record or paper)(IHIS)
   * Foley catheter
   * Video of echocardiogram of normal heart (transesophageal four chamber and transgastric short axis)
   * Alaris pump for delivery for IV anesthetics (Epinephrine, Nitroprusside, and Insulin) Learner Information (Information given to learner during scenario)

   Scenario Introduction (give to learner in all 3 scenarios):

   Your patient is a 57 year old male who is undergoing a triple vessel CABG (LIMA to LAD, saphenous to RCA, and saphenous to OM). In addition to CAD the patient has a history of type 2 DM and HLD. The surgeon has completed the last graft with a total bypass time of 45 minutes. The procedure has been uncomplicated to this point. The patient has an arterial line, a 16 g IV, and an introducer with a PAC. The patient is on no infusions and is receiving isoflurance via the bypass machine. The patient is currently paralyzed. There is transesophageal echocardiogram available. The surgeon has placed epicardial pacing wires. Your task will be to wean the patient off of CPB.

   General Information (SBAR):

   Name: Jerry Gergich Age: 57 Birth Date: 10/28/1957 Weight: 90 kg Height: 5'10'' Vital Signs: HR 65 (sinus), BP 122/80, RR 14, SpO2 98%

   Patient History:

   History of Present Illness: unstable angina x 1 month Allergies: NKDA Medications: carvedilol, glyburide, aspirin Past Medical / Surgical History: inguinal hernia repair (uneventful GA) Intake/outputs: n/a

   Symptoms:

   Events leading up to Illness: worsening chest pain Onset of symptoms: 1 month Provocation / provokes: exertion Severity of pain: 5/10 Review of Systems CNS: AAO x 3, no neurologic deficits Cardiovascular: chest discomfort with exertion, no syncope or dyspnea Pulmonary: normal; no wheezing, cough Abdominal: within normal limits

   Physical Exam:

   Airway: MP 2, good neck extention, normal TM distance, good oral opening Chest: RRR, no murmurs; lungs clear Abdominal: within normal limits Neuro: within normal limits

   Laboratory, Radiology, and Other Relevant Studies: Labs:
   * Labs: Hct 39, platelets 360 on admission
   * Chemistry: within normal limits
   * Type and Cross: negative antibody screen; 4 units available
   * PT, PTT, INR: within normal limits
   * LHC: 90% stenosis of LCA, RCA and OM.
   * Echo: Normal LV and RV size and function; LV EF 55%
   * EKG: NSR, Inverted T waves in leads II and V5.

   Simulation Sequence

<!-- -->

1. On Bypass

   Vital signs:

   HR BP SPO2 RR ETCO2 CVP PAP CO Temp 40 50 100 n/a n/a 5 5/3 n/a 35

   EKG: junctional bradycardia Appearance/PE: intubated, sedated, paralyzed, on CPB Operator details: After receiving hand-off the surgeon will announce that he will soon be removing the aortic cross-clamp.

   Learner Objectives and Interventions: The participant should make sure he/she receives a thorough hand-off with a clear understanding of the patient's background and surgical course. The resident should call his/her attending physician in preparation for weaning from CPB.

   Transition Cue: Removal of Cross Calmp Go to state: Maintenance
2. Ventricular Fibrillation

   Vital signs:

   HR BP SPO2 RR ETCO2 CVP PAP CO Temp n/a 40 100% n/a n/a 4 5/2 n/a 35.3

   EKG: Ventricular fibrillation Appearance/PE: anesthetized, paralyzed, on CPB Operator details: Surgeon will continue to operate without noticing the rhythm. If the participant does not recognize the rhythm within 30 seconds the perfusionist will announce that he is giving 100 mg lidocaine via the bypass machine.

   Learner Objectives and Interventions: The participant should recognize the arrhythmia and direct the surgeon to administer shocks to the patient.

   Transition Cue: Defibrillation Go to state: Junctional Bradycardia
3. Junctional Bradycardia

   Vital signs:

   HR BP SPO2 RR ETCO2 CVP PAP CO Temp 40 50 100 n/a n/a 4 5/2 n/a 35.3

   EKG: junctional bradycardia Appearance/PE: Anesthetized, paralyzed, on CPB Operator details: The surgeon will ask for the participant to begin ventilating the patient.

   Learner Objectives and Interventions: Participant should ventilate the patient with adequate tidal volumes/rate. Ask for pacer box and begin pacing the patient. If the participant does not ask for it, the perfusionist will simply bring the participant a pacing box (pre-set to 80; v-paced)

   Transition Cue: Pacing Go to state: Hyperkalemia
4. Hyperkalemia

Vital signs:

HR BP SPO2 RR ETCO2 CVP PAP CO Temp 80 50 100 Vent 20 5 4/2 n/a 35.7

EKG: V-paced Appearance/PE: Anesthetized, paralyzed, mechanically ventilated, on CPB Operator details: If the participant has not already asked for it at this point, the perfusionist will bring him/her the results for an ABG: (pH 7.4, paO2 350, paCO2 34, HCO3 22, K+ 6, Glu 250, Ca++ 4, Hct 24). The surgeon will ask if he can come off of bypass.

Learner Objectives and Interventions: The participant should treat the underlying metabolic disturbance (mainly hyperkalemia and hyperglycemia) before allowing the surgeon to proceed with removal from bypass. If insulin is given the patient will progress to state: "wean off". If no insulin is given the patient will go back to state 2: "ventricular fibrillation".

Transition Cue: Insulin Given Go to state: Wean Off

Transition Cue: Insulin Not Given Go to state: Ventricular Fibrillation

4. Wean Off

Vital signs:

HR BP SPO2 RR ETCO2 CVP PAP CO Temp 80 78/50 100 Vent 22 6 5/2 n/a 35.8

EKG: V-paced Appearance/PE: Anesthetized, paralyzed, mechanically ventilated, on CPB Operator details: Surgeon will ask which drips the patient is on. Learner Objectives and Interventions: The participant should look at the echocardiogram (which will reveal a normal heart). The participant should provide inotropic support (low dose epinephrine drip) at which point the BP will increase to approximately 110/60 over 30 seconds. The scenario will then end.

The Ohio State University CSEAC 2nd Scenario Development Form Scenario Name: Protamine Reaction Content expert: Sujatha Bhandary MD Date of Development: 8/29/14 Targeted Audience: CA-2, CA-3 anesthesia residents Simulation Platform: HPS

*Synopsis of Scenario:

The purpose of this scenario is to expose trainees to a severe type III protamine reaction after weaning off of cardiopulmonary bypass. Although the most severe reaction to administration of protamine (severe pulmonary vasoconstriction, RV failure, systemic hypotesnsion) is rare, the result can be catastrophic. High fidelity simulation provides an opportunity for trainees to get exposure to this entity in a safe, controlled environment. The scenario will be followed by both a debriefing session to allow the participants to reflect on their performance and a short didactic session on proper administration of protamine and the pathophysiology of protamine reactions.

The scenario will begin after completion of the previous scenario: "Weaning from Cardiopulmonary Bypass". As before the patient is a 57 year old male who has just undergone an uncomplicated triple vessel CABG with 45 minutes of bypass time. The patient was successfully weaned off of CPB after treatment of hyperkalemia (see prior scenario). This scenario can begin either after debriefing the previous scenario or may begin without interruption. The surgeon will start the scenario by asking the participant to administer protamine. At this point the patient is hemodynamically stable (V-paced at 80, BP 110/60, PAP 30/15, CO 5.2). The patient will start the scenario on an epinephrine drip at 0.02 mcg/kg/min. The participant will be informed that the patient was given 30,000 unites of heparin in preparation for going on CPB. The last ACT was 468. The patient will not have any hemodynamic changes in response to a test dose of protamine, and the participant should continue to administer the appropriate dose. After 2 minutes without a change in vitals the patient will begin to undergo hemodynamic changes consistent with a type III protamine reaction over the course of 5 minutes (hypotesnsion, desaturation, decreased cardiac output, pulmonary hypertension). Upon recognizing the problem the participant should discontinue the protamine infusion, call for help, communicate with the surgeon, and provide supportive care for the patient. An echocardiogram (upon request) will demonstrate a dilated RV. Intervening to stop the protamine and administer vasopressors will stabilize the patient, however failure to act will result in cardiovascular collapse and necessitate going back on CPB.

Learning Objectives:

5.Demonstrate appropriate administration of protamine following cardiopulmonary bypass.

6.Recognize the signs of an acute type III protamine reaction and respond appropriately.

7.Describe the different types of protamine reactions, the pathophysiology of each, and the risk factors for developing them.

Scenario Intro (read to learner) Your patient is a 57 year old male who is undergoing a triple vessel CABG (LIMA to LAD, saphenous to RCA, and saphenous to OM). In addition to CAD the patient has a history of type 2 DM and HLD. The procedure has been uncomplicated to this point. The patient has an arterial line, a 16 g IV, and an introducer with a PAC. The patient is currently paralyzed. There is a transesophageal echocardiogram available upon request. The patient as already been successfully weaned off of CPB and is hemodynamically stable on a low dose epinephrine drip.

*Facilitator briefing/ Curricular information: Prior to receiving hand-off and beginning the scenario the participant will be handed a sheet with the patient's pre-op history and physical already completed. All labs and imaging will be provided. The resident will have the opportunity to ask additional questions to the departing provider. The confederates in the room will include the cardiac surgeon and a perfusionist. Echocardiography will be available upon request as will arterial blood gases. The patient will already be on an epinephrine infusion at 0.02 mcg/kg/min. Other cardiac drugs (lidocaine, amiodarone, nitroglycerine, norepinephrine, vasopressin) will be drawn up and available. Epicardial wires coming from the surgical field will be connected to a pacing box set at 80 (V-paced).

Educational Learning Model

Prerequisites: Completion of cardiac anesthesiology rotation Didactics Needs: Powerpoint presentation, debriefing room Learning Method: Experiential Debriefing Method: Guided reflection with peer feedback. Didactic content.

Preparation Supporting Files

* Patient preoperative report
* PowerPoint presentation

Roles

* Cardiac Surgeon
* Perfusionist

Setting

* OR
* Patient intubated, sedated, paralyzed, on CPB

Monitors Available to Participant • Code Cart with pacing/defibrillation pads

* EKG monitoring
* Five-lead electrocardiogram
* Pulse-oximetry
* Temperature probe
* Capnography
* Arterial catheter
* Central venous catheter
* Pulmonary artery catheter
* Transesophageal Echocardiogram

Other Equipment Required

• Anesthesia machine that has passed the check out

* Airway equipment on the cart including Macintosh 3 and Miller 2 blades, endotracheal tube sizes 6 and 7 with stylet and empty 10 mL syringe
* Two prepared 1000 mL intravenous fluid bags on blood infusion lines
* Pharmacologic agents available upon request: propofol, etomidate, ketamine, succinylcholine, vecuronium, midazolam, fentanyl, atropine, ephedrine, phenylephrine, epinephrine (in syringe and prepared in 100 mL saline bag), norepinephrine (in syringe and prepared in 100 mL saline bag), vasopressin, neostigmine, glycopyrrolate, metoprolol, esmolol,
* Epinephrine, Nitroprusside, and Insulin drips connected to a manifold and in line with the patient's CVC
* Yankauer suction
* Record keeping material (compurecord or paper)(IHIS)
* Foley catheter
* Video of echocardiogram of normal heart (transesophageal four chamber and transgastric short axis)
* Alaris pump for delivery for IV anesthetics (Epinephrine, Nitroprusside, and Insulin)
* Pacing Box Learner Information (Information given to learner during scenario)

  1. Initial Baseline

     Vital signs:

     HR BP SPO2 RR ETCO2 CVP PAP CO Temp 80 110/60 100 Vent (14) 30 12 30/15 5.4 36 EKG: V-paced Appearance/PE: intubated, sedated, paralyzed, on vent Operator details: Epi infusion running at 0.02 mcg/kg/min into patient's central line. This scenario state will take off directly after the final state of the prior scenario ("weaning off CPB"). The surgeon will ask for protamine to be given. If the participant asks the perfusionist will inform him/her that the total heparin dose was 30,000 units and the last ACT was 468. The test dose will be negative (no change in vital signs).

     ABG (if requested): pH 7.34, PaO2 350, PaCO2 35, HCO3 23, K+ 4.4, Ca++ 4, Glu 180, Hct 23) Learner Objectives and Interventions: Calculation of proper reversal dose of protamine. Administration of test dose of protamine and slow administration of full reversal dose with careful attention to potential hemodynamic changes.

     Transition Cue: Administration of Protamine Go to state: Protamine Reaction
  2. Protamine Reaction

     Vital signs:

     HR BP SPO2 RR ETCO2 CVP PAP CO Temp 80 70/35 92% Vent (14) 20 28 60/45 36 EKG: V-pace Appearance/PE: anesthetized, paralyzed, on vent Operator details: Changes in vital signs will occur slowly (over 5 minutes). Surgeon will continue to operate without noticing the changes in vital signs. An Echo (if requested) will show a dilated RV. Stopping the infusion and administration of vasopressors will result in stabilization. Failure to stop the infusion will lead to further deterioration.

     Learner Objectives and Interventions: Discontinue protamine infusion. Communicate with surgeon. Call for help. Provide supportive care for the patient (vasopressors).

     Transition Cue: Stop Infusion Go to state: Stabilization Transition Cue: Failure to Stop Infusion Go to state: Severe Reaction
  3. Stabilization

     Vital signs:

     HR BP SPO2 RR ETCO2 CVP PAP CO Temp 80 95/57 95 Vent (14) 30 16 40/20 36 EKG: V-paced Appearance/PE: intubated, sedated, paralyzed, on vent Operator details: Vitals will stabilize to current state over 2 minutes following discontinuation of protamine and administration of vasopressors. Surgeon will ask if the provider can restart the protamine now. After discussion with surgeon the scenario will end.

     Learner Objectives and Interventions: Discuss with surgeon options for reversal of heparin.
  4. Severe Reaction

Vital signs:

HR BP SPO2 RR ETCO2 CVP PAP CO Temp 80 45/20 89 Vent (14) 15 23 70/44 36

EKG: V-paced Appearance/PE: intubated, sedated, paralyzed, on vent Operator details: Failure to stop the infusion will result in worsening of the patient's condition to the current state. Surgeon will now became aware of the hemodynamic changes and will insist on going emergently back on CPB. The scenario will end.

The Ohio State University CSEAC 3rd Scenario Development Form Scenario Name: Coronary Air After Bypass Grafting Content expert: Sujatha Bhandary MD Date of Development: 8/29/14 Targeted Audience: CA-2, CA-3 anesthesia residents Simulation Platform: HPS

Synopsis of Scenario:

The purpose of this scenario is for the participant to take a thoughtful, systematic approach to the sudden onset of ST changes and hypotension following completion of coronary artery bypass graft (CABG) surgery. Specifically this scenario will deal with intracoronary air, which if unrecognized can be fatal. Residual air has been reported to be present as in as much as 12% of patients undergoing CABG surgery.* This simulation will give residents the chance to treat this condition in a safe, constructive environment so that they will be more comfortable with diagnosing this rare but potentially devastating condition. The simulation is intended to rely on the residents' knowledge of cardiac physiology, and basic echocardiography interpretation.

The scenario will start following the completion of the previous scenario (Protamine Reaction) at which the time patient has been successfully weaned off of bypass and the chest has just been closed. Immediately after beginning the scenario the surgeon will leave the room. At this time the fellow (confederate) will begin to suture the skin. Shortly thereafter the patient will have ST elevation in the inferior EKG leads. The fellow will ask if the echocardiogram looks okay. A mid-esophageal four-chamber view of the patient's heart will demonstrate air bubbles in the left ventricle. A trans-gastric short axis view of the heart (if requested) will show the inferior wall of the heart to be akinetic. The patient will become hypotensive with decreased cardiac index. The resident should simultaneously form a differential diagnosis and treat the symptoms while communicating to the surgeon his/her findings. Ultimately the resident should request that the surgeon reopen the patient's chest and purge the intra-cardiac air. Failing to do so will result in the patient going into cardiogenic shock and ventricular fibrillation.

Learning Objectives:

8. Form a differential for post CABG hypotension and EKG changes. 9. Diagnose intra-cardiac air and regional wall motion abnormalities on echocardiogram.

10. Effectively treat cardiogenic shock with pharmacologic agents. 11. Communicate with the surgeon regarding the need for surgical intervention.

Scenario Intro (read to learner) Your patient is a 57 year old male who is undergoing a triple vessel CABG (LIMA to LAD, saphenous to RCA, and saphenous to OM). In addition to CAD the patient has a history of type 2 DM and HLD. The surgeon completed the grafts with a total bypass time of 45 minutes. The patient has been weaned of cardiac bypass and successfully reversed with protamine. The chest has just been closed. The procedure has been uncomplicated to this point. The patient has an arterial line, a 16 g IV, and an introducer with a PAC. The patient is on a low dose epinephrine infusion (.0.02 mcg/kg/min). The patient is currently paralyzed. There is a transesophageal echocardiogram available upon request. The surgeon has placed epicardial pacing wires. You will be responsible for transitioning the patient to the cardiac ICU.

Facilitator briefing/ Curricular information:

Prior to receiving hand-off and beginning the scenario the participant will be handed a sheet with the patient's pre-op history and physical already completed. All labs and imaging will be provided. The resident will have the opportunity to ask additional questions to the departing provider. The confederates in the room will include the cardiac surgeon and a perfusionist. Echocardiography will be available upon request as will arterial blood gases. The patient is on a low dose epinephrine infusion (0.02 mcg/kg/min). Other cardiac drugs (lidocaine, amiodarone, nitroglycerine, norepinephrine, vasopressin) will be drawn up and available. Epicardial wires coming from the surgical field. These can be connected to a pacing box which will provided upon request.

Educational Learning Model Prerequisites: Completion of cardiac anesthesiology rotation Didactics Needs: Powerpoint presentation, debriefing room Learning Method: Experiential Debriefing Method: Guided reflection with peer feedback. Didactic content. Preparation Supporting Files • Patient preoperative report

* PowerPoint presentation Roles
* Cardiac Surgeon
* Perfusionist Setting
* OR
* Patient intubated, sedated, paralyzed, on CPB

Monitors Available to Participant • Code Cart with pacing/defibrillation pads • EKG monitoring • Five-lead electrocardiogram • Pulse-oximetry

• Temperature probe

* Capnography
* Arterial catheter
* Central venous catheter
* Pulmonary artery catheter
* Transesophageal Echocardiogram

Other Equipment Required • Anesthesia machine that has passed the check out

• Airway equipment on the cart including Macintosh 3 and Miller 2 blades, endotracheal tube sizes 6 and 7 with stylet and empty 10 mL syringe

• Two prepared 1000 mL intravenous fluid bags on blood infusion lines

• Pharmacologic agents available upon request: propofol, etomidate, ketamine, succinylcholine, vecuronium, midazolam, fentanyl, atropine, ephedrine, phenylephrine, epinephrine (in syringe and prepared in 100 mL saline bag), norepinephrine (in syringe and prepared in 100 mL saline bag), vasopressin, neostigmine, glycopyrrolate, metoprolol, esmolol,

* Epinephrine, Nitroprusside, and Insulin drips connected to a manifold and in line with the patient's CVC
* Yankauer suction
* Record keeping material (compurecord or paper)(IHIS)
* Foley catheter
* Video of echocardiogram 2 views (transesophageal four chamber with intracardiac air in LV and transgastric short axis with akinetic inferior wall)
* Alaris pump for delivery for IV anesthetics (Epinephrine, Nitroprusside, and Insulin

  *Learner Information (Information given to learner during scenario)

Simulation Sequence

1. Chest Closed

   Vital signs:

   HR BP SPO2 RR ETCO2 CVP PAP CO Temp 70 110/60 100 14 (vent) 35 12 30/15 5 36.3

   EKG: normal sinus rhythm Appearance/PE: intubated, sedated, paralyzed; chest closed Operator details: The surgeon has just finished closing the chest at which time he/she will give a sign out and leave the room.

   Learner Objectives and Interventions: The participant should make sure he/she receives a thorough hand-off with a clear understanding of the patient's background and surgical course.

   Transition Cue: Surgeon leaves the room Go to state: ST elevation
2. ST Changes

   Vital signs:

   HR BP SPO2 RR ETCO2 CVP PAP CO Temp 70 110/60 100% 14 (vent) 35 12 30/15 5 36.3

   EKG: Normal sinus rhythm; ST depression in AVF, II, III Appearance/PE: intubated, sedated, paralyzed; chest closed Operator details: Fellow will begin suturing the skin and will ask the participant what the cardiac index is. At this point the patient should experience ST depression in the inferior leads.

   Learner Objectives and Interventions: The participant should recognize the EKG changes and look to the echocardiogram for clinical correlation. He/She should communicate with the surgical team.

   Transition Cue: Learner looks at Echocardiogram Go to state: ST Elevation
3. ST Elevation

   Vital signs:

   HR BP SPO2 RR ETCO2 CVP PAP CO Temp 70 85/50 100 14 (vent) 27 10 40/25 1.5 36.3

   EKG: normal sinus rhythm; ST elevation in AVF, II, III Appearance/PE: Intubated, sedated, paralyzed; chest closed Operator details: TEE four chamber view will demonstrate air bubbles in the LV. Trans-gastric short axis will show akinetic inferior wall. Patient will get hypotensive over 2 minutes, but will responds to IV epinephrine.

   Learner Objectives and Interventions: Participant should form differential for hypotention with ST elevation, and treat pharmacologically with epinephrine. The participant should communicate with the surgeon regarding the need for re-opening at which point the scenario will end. If he/she does not communicate with the surgical team the patient will decompensate and go into VFib.

   Transition Cue: Failure to communicate with surgeon Go to state: VFib
4. VFib

Vital signs:

HR BP SPO2 RR ETCO2 CVP PAP CO Temp n/a - - 14 (vent) 0 0 0 0 36.3

EKG: V-fib Appearance/PE: Intubated, sedated, paralyzed; chest closed Operator details: Failure to communicate with the team regarding intracardiac air and need to re-open will result in worsening cardiogenic shock developing to ventricular fibrillation. Surgeon will re-enter room and ask what happened.

Learner Objectives and Interventions: Recognize ventricular fibrillation and begin ACLS (epinephrine/defibrillation). Regonize intracoronary air as ca

ELIGIBILITY:
Inclusion Criteria:

* Resident physicians who have completed at least one month of cardiac rotation are included.This high fidelity simulation lab course if offerred to every resident that meets the criteria.This is a part of their educational activity.At the beginning of the course they are given the option to participate in the survey.If they do not wish to participate in the survey it will not affect their education.Participitaion in the survey is purely voluntary.

Exclusion Criteria:

* Resident physicians that did not wish to participate in filling out the survey or not able to fill out the survey.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Resident physicians who have completed at least one month of cardiac rotation are included.This high fidelity simulation lab course if offered to every resident that meets the criteria.This is a part of their educational activity.At the beginning of the course they are given the option to participate in the survey.If they do not wish to participate in the survey it will not affect their education.Participation in the survey is purely voluntary.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
Use of NASA Task Load Index Scale in the Evaluation of Neuro-Cognitive Workload during Cardiac Anesthesia Based Simulation Scenarios | 2 years
  The NASA-TLX Scale is a multi-dimensional tool used to evaluate subjective workload in subjects performing a task. The scale uses six factors to evaluate the magnitude and source of the workload in human subjects with both high reliability and sensitivity. The scale has been one of the gold standards for cognitive workload measure for over thirty years.

CONTACTS AND LOCATIONS:
Overall Officials: Sujatha P Bhandary, M.D., Principal Investigator — Ohio State University